CLINICAL TRIAL: NCT04390724
Title: Yttrium-90 Radiation Lobectomy: Dose Optimization and Prediction of FLR Hypertrophy to Enable Resection of HCC
Brief Title: Optimizing Y90 Therapy for Radiation Lobectomy
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert Lewandowski, Professor of Radiology, Medicine, and Surgery, Northwestern University
Other Study IDs: STU00209629
Record Dates: First submitted 2020-05-11; First posted 2020-05-15 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: HCC; Resection; Transplant; Metastatic Cancer; Adult Primary Liver Cancer
Keywords: HCC; Y90 Radioembolization; Liver Resection; Liver Transplant; Liver Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Group 1 patients consent to have an optional study-specific liver parenchymal biopsy Group 2 have their blood drawn to measure circulating trophic factors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Patient Group 1: Y90 Standard-of-Care: The first group of patients will be treated with Y90 dose and embolic load as per standard-of-care
  Interventions: Device: Y90 radioembolization
- Patient Group 2: Y90 Dose determined by results from Group 1: The second group of patients will be treated with the optimal Y90 dose and embolic load found in Patient Group 1
  Interventions: Device: Y90 radioembolization

INTERVENTIONS:
Device: Y90 radioembolization — Patients with HCC who are eligible to receive standard-of-care Y90 radioembolization and are hepatic resection candidates with inadequate future liver remnant
  Other Names: Patient Group 1: Y90 Standard-of-Care; Patient Group 2: Y90 Dose determined by results from Group 1

SUMMARY:
HCC resection candidates with inadequate future liver remnant will be enrolled in this study. They will be treated with Y90 radioembolization to help grow the liver enough to undergo liver resection. There will be 2 Patient Groups. The first group of patients will be treated with Y90 dose and embolic load as per standard-of-care. The second group of patients will be treated with the optimal Y90 dose and embolic load found in Patient Group 1.

DETAILED DESCRIPTION:
In this study there will be 2 different patient groups 1 and 2 that will consist of 40 and 64 patients, respectively with hepatocellular carcinoma who are eligible for resection and to receive Y90 radioembolization who have inadequate future liver remnant.

Y90 radioembolization uses radioactive beads (microspheres), which are tiny glass particles that are loaded with radiation. The beads are injected into an artery of the liver that supplies blood to the tumor(s). The beads flow to the tumor(s) and become trapped inside. The beads release the Y90 radiation inside the tumor(s).

Liver resection is used to remove the part of the liver that has the HCC tumor(s). It has been shown that Y90 radioembolization can also increase the untreated liver's size and volume. Patients with HCC may be liver resection candidates if they have a large enough liver.

The purpose of this research is to determine if there is an ideal Y90 dose to increase liver volume of the future liver remnant. This research may help determine the best Y90 dose for future patients who need a larger liver to have a liver resection.

Participants in Group 1 will have standard-of-care Y90 radioembolization as well as study-specific optional liver biopsy.

Participants who already have a planned Y90 radioembolization treatment with the dose range established in Group 1 will be enrolled into Group 2. Patient Group 2 will have blood drawn and a quantitative MRI performed at specific timepoints.

The study will last up to 3 months. Participants' health status will be followed up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have been diagnosed with HCC confirmed by histology or must meet one of the following American Association for the Study of Liver Diseases (AASLD) guidelines:

   * AFP >200 and radiological evidence (arterial hypervascularity) of lesion > 2 cm does not require biopsy
   * Two imaging modalities (triphasic CT, MRI, ultrasound, angiography) demonstrating arterial hypervascularity in the background of cirrhosis does not require biopsy
   * One imaging modality with a lesion with arterial hypervascularity with wash out in early or delayed venous phase, does not require a biopsy
2. Child-Pugh stage A
3. Future Liver Remnant (FLR) of < 40%
4. ECOG Performance Status 0-1
5. Bilirubin ≤ 3.0 mg/dl- Treatment may proceed if the Bilirubin is elevated if the tumor may be isolated from a vascular standpoint
6. Creatinine ≤ 2.0 mg/dl
7. ANC ≥ 1.5 K/uL
8. Platelets > 25 K/uL
9. Patient is willing participate in this study and has signed the consent
10. For Group 2 patients only:

    * Patients planned Y90 dose and embolic load is found to fall within the optimal dose and embolic load size from data from Group 1 patients

Exclusion Criteria:

1. Patient must not be pregnant

   NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy
   * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
2. For Patients in Group 2 only:

   * Patients who have contraindications to MRI:

     * Patients that are claustrophobic and haven't been able to tolerate an MRI in the past. (Patients with mild claustrophobia are eligible and have the option to take

       1mg oral Lorazepam prior to the MRI, if needed)
     * Allergy to gadolinium-containing contrast media
     * Patients with a pacemaker, metallic clip, aneurysm clips, shrapnel fragments, etc.
     * Patients with an eGFR < 30 mL/min/m²
3. Must not have any significant life-threatening extra-hepatic disease or life- threatening secondary malignancies, including patients who are on dialysis, have unresolved diarrhea, have serious unresolved infections including patients who are known to be HIV positive or have acute HBV or HCV
4. Must not have any contraindications to angiography and selective visceral catheterization such as bleeding diathesis or coagulopathy that is not correctable by usual therapy of hemostatic agents (e.g. closure device)
5. Must not have any co-morbid disease or condition that would place the patient at undue risk and preclude safe use of TheraSphere treatment, in the Investigator's judgment
6. History of severe peripheral allergy or intolerance to contrast agents, narcotics, sedatives or atropine that cannot be managed medically

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years and older with HCC who are eligible to receive standard-of-care Y90 radioembolization and are hepatic resection candidates with inadequate future liver remnant
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Patient Group 1: Y90 Glass Microspheres | 2 years
  Measure the distribution of Y90 glass microspheres throughout the tumor and non-tumor hepatic parenchyma, as assessed by same day post-radioembolization study-specific non-FDG PET/CT scan.
Patient Group 1: Sphere distribution | 2 years
  Sphere distribution will be correlated with mean lobar absorbed radiation dose, embolic load, and time taken to achieve adequate Future Liver Remnant (>40% of total liver volume) to determine optimal lobar dose and embolic load.
Patient Group 2: Quantitative Imaging Radiologic Biomarkers | 3 years
  Quantitative MRIs and biomarkers drawn will assess the association of circulating and imaging biomarkers on Future Liver Remnant hypertrophy. Tropic factor biomarkers to be drawn include: hepatocyte growth factor, epidermal growth factor, transforming growth factor beta, interleukin-6, tumor necrosis factor alpha, insulin-like growth factor binding protein, vascular endothelial growth factor, platelet derived growth factor, and phosphorus level.
Patient Group 2: HCC Resection | 3 years
  Assess progression-free survival between patients with HCC who underwent resection following Y90 radioembolization and those who presented with an adequate Future Liver Remnant for resection (i.e. who were not treated pre-surgically).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lewandowski, MD, Principal Investigator — Northwestern University; Jeremy Collins, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No